CLINICAL TRIAL: NCT07174856
Title: The Misoprostol-Only Regimen Evidence (MORE) Study: A Randomized Controlled Trial Comparing the Misoprostol-only Regimen Versus the Combined Mifepristone and Misoprostol Regimen for Medication Abortion
Brief Title: The Misoprostol-Only Regimen Evidence Study
Acronym: MORE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ibis Reproductive Health (Other)
Collaborators: University of Utah (Other); Planned Parenthood Association of Utah (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1394391
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Abortion, Medical
Keywords: misoprostol; mifepristone; medication abortion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Combined regimen (Active Comparator): Participants in this arm are randomized to receive the standard of care combined mifepristone + misoprostol regimen. Specifically, for those with pregnancies <64 days, mifepristone (200mg orally) followed 24-48 hours later by misoprostol (800μg b/v); for those 64-77 days, they will take a second dose of misoprostol (800μg b/v) taken 3 hours later.
  Interventions: Drug: Combined regimen
- Misoprostol-only (Experimental): Participants in this arm will be randomized to receive a misoprostol-only regimen. Specifically, 3-4 doses of 800μg misoprostol administered sublingually every 3 hours.
  Interventions: Drug: Misoprostol-only medication abortion regimen

INTERVENTIONS:
Drug: Misoprostol-only medication abortion regimen — This intervention is an updated misoprostol-only regimen that involves being counseled on and receiving medications for a medication abortion using 3-4 doses of 800μg misoprostol administered sublingually every 3 hours.
  Arms: Misoprostol-only
Drug: Combined regimen — This intervention will involve participants being counseled on and receiving medications for a medication abortion regimen of mifepristone (200mg orally) followed 24-48 hours later by misoprostol (800μg b/v) with a second dose of misoprostol (800μg b/v) taken 3 hours later only for those 64-77 days.
  Arms: Combined regimen

SUMMARY:
The goal of this study is to evaluate the effectiveness, non-inferiority, and side-effect profile of an updated misoprostol-only regimen, as compared to the combined mifepristone-misoprostol regimen, among people seeking medication abortion (MAB) through 77 days of pregnancy in telehealth and in-person settings. The investigators aim to evaluate this in both in-clinic and telehealth medication abortion care in the United States.

The main questions it aims to answer are:

1. What proportion of pregnant people using an updated misoprostol-only medication abortion regimen have a complete abortion using just the prescribed pills?
2. Is the updated misoprostol-only medication abortion regimen no more than 5% less effective (non-inferior) than the standard combined medication abortion regimen?
3. What is the pattern of beta hCG decline following use of a misoprostol-only medication abortion through 77 days of pregnancy?

Participants will:

* be randomized to one of two medication regimens (misoprostol-only or the combined regimen) in a 1:1 ratio based on duration of pregnancy at enrollment. - self-report outcomes via daily surveys for the first 3 days, and thereafter weekly at 7, 14, 21, 28, and 35 days.
* return to the clinical site for tests as instructed

The investigators hypothesize that the proportion with complete abortions in the misoprostol-only arm will be non-inferior to the proportion with complete abortions in the combined regimen arm within a 5% margin of inferiority

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing misoprostol-only (3-4 doses x 800μg misoprostol sublingually every 3 hours) (Arm 2) to the combined regimen (<64 days: mifepristone (200mg orally) followed 24-48 hours later by misoprostol (800μg b/v) with a second dose of misoprostol (800μg b/v) taken 3 hours later only for those 64-77 days) (Arm 1). The combined regimen is the standard of care for medication abortion in the United States, and both regimens are widely used across the globe for termination of pregnancy. Participants will be randomized to each group in a 1:1 ratio based on duration of pregnancy at enrollment. The primary outcome is the proportion who have a complete abortion (no ongoing pregnancy) without procedural intervention or additional doses of medication as determined by negative HSPT between 28-42 days, ultrasound, or declining serum beta hCG by clinic protocols. Side effects, additional interventions, adverse events, acceptability, and quality of care will be assessed with daily surveys for the first 3 days, and thereafter weekly at 7, 14, 21, 28, and 35 days.

The primary outcome for this study is complete abortion, defined as successful expulsion of the intrauterine pregnancy without need for procedural intervention or additional doses of medication during the follow-up period as determined by negative HSPT between 28-42 days, ultrasound, or declining serum beta hCG by clinic protocols. The investigators will report abortion completion overall by study arm. Additionally, the investigators will evaluate and report on the non-inferiority of abortion completion following use of the misoprostol-only regimen as compared to the combined mifepristone and misoprostol regimen.

Participants will be determined to have had a complete abortion without need for procedural intervention or additional doses of medication, and the investigators will also report the number and proportion of complete abortions as defined more broadly by the MARE guidelines as successful expulsion of the intrauterine pregnancy without need for procedural intervention.

Secondary study endpoints include:

• change in serum beta hCG 7-14 days following use of the misoprostol-only regimen and in the mifepristone-misoprostol regimen

In more detail, secondary outcomes to be measured include declines in serum beta hCG between baseline and 7-14 days among a subset of participants to characterize patterns following use of the misoprostol-only regimen and the combined mifepristone-misoprostol regimen.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy of < or = 77 days duration based on LMP or ultrasound
* Positive pregnancy test (self-report or in-clinic)
* Age: States without parental involvement laws : in-person patients ages 14 years and older; States with parental involvement or notification laws: 18 years or older
* Willing and able to give informed consent
* Willing to comply with study protocol
* Willing to record requested information in the study surveys
* English or Spanish speaking
* Has a text message, email, or phone call capable device for survey completion
* Understands and signs an Institutional Review Board (IRB) approved informed consent form prior to undergoing any study procedures or randomization

Exclusion Criteria:

* concurrent participation in any other interventional trial
* unwilling to comply with the study protocol and survey/visit schedule
* contraindication to mifepristone (chronic corticosteroid administration, adrenal disease)
* contraindication to misoprostol (glaucoma, mitral stenosis, sickle cell anemia, or known allergy to prostaglandin)
* cardiovascular disease (angina, valvular disease, arrhythmia, or cardiac failure)
* diagnosis of porphyria
* known bleeding disorder or receiving anticoagulants
* pregnancy with an IUD in place
* diagnosis of pregnancy of unknown location (PUL), early pregnancy failure, incomplete or inevitable abortion (absent gestational sac and/or open cervical os)
* possibility of ectopic pregnancy
* known or suspected pelvic infection
* Have issues or concerns (in the judgement of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.
* Have previously participated in the study
* Be a site staff member with delegated study responsibilities or a family member of, or have a close relationship with, a site staff member with delegated study responsibilities.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Abortion completion | 28-42 days after taking the pills
  The primary outcome for this study is complete abortion, defined as successful expulsion of the intrauterine pregnancy without need for procedural intervention or additional doses of medication during the follow-up period as determined by negative HSPT, ultrasound, or declining serum beta hCG by clinic protocols.
Non-inferiority of the misoprostol-only regimen | Completion measured 28-42 days after taking the pills
  Study investigators will evaluate and report on the non-inferiority of abortion completion following use of the misoprostol-only regimen as compared to the combined mifepristone and misoprostol regimen within a 5% margin of inferiority.

SECONDARY OUTCOMES:
hCG decline | Change in beta hCG between 0 and 7-14 days post medication abortion
  We will measure declines in serum beta hCG between baseline and 7-14 days among a subset of participants to characterize patterns following use of the misoprostol-only regimen and the combined mifepristone-misoprostol regimen.

CONTACTS AND LOCATIONS:
Locations (1):
- Planned Parenthood Association of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share a de-identified dataset that includes at a minimum: treatment group, adherence to treatment, and primary outcome (abortion completion).
Supporting Information: Study Protocol
Time Frame: At a minimum, we will make key components of the study protocol as well as a de-identified dataset with key data elements available to members of the scientific community within 6 months of publication of the primary and secondary study outcomes.
Access Criteria: Interested researchers can contact the study team with a brief analysis plan and the research team will share the data with those researchers.